CLINICAL TRIAL: NCT02754466
Title: Oral Health and Its Relation to Growth, Development and Well-being of Schoolchildren Before and After Restorative Treatments
Brief Title: Oral Health and Its Relation to Development and Well-being of Schoolchildren Before and After Restorative Treatments
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Children could not be examined longer than 2 years due to COVID-19 pandemic and schools closure.
Sponsor: University of Brasilia (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Leandro Hilgert, Professor of Operative Dentistry, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.400.687/2016
Record Dates: First submitted 2016-04-18; First posted 2016-04-28 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Dental Caries; Dental Atraumatic Restorative Treatment; Oral Health
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep dentin lesions (Experimental): Subjective vs objective criteria in selective excavation of carious lesions Group 1: selective carious dentin excavation using subjective criteria (standard protocol in Dentistry) Group 2: selective carious dentin excavation using objective criteria (polymer burs) All restorations performed using high-viscosity glass-ionomer.
  Interventions: Other: Subjective vs objective criteria in selective excavation
- Shallow and medium depth dentin lesion (Experimental): Glass-ionomer vs Bulk fill composites in the ART approach All cavities excavated using hand-instruments only (ART approach) Group 1: restorations using high-viscosity glass-ionomer Group 2: restorations using self-etch adhesive and bulk fill composite
  Interventions: Other: Glass-ionomer vs Bulk fill composites in the ART approach

INTERVENTIONS:
Other: Subjective vs objective criteria in selective excavation — Subjective vs Objective criteria (Polymer burs) to perform selective excavation of dentin caries in deep lesions
  Arms: Deep dentin lesions
Other: Glass-ionomer vs Bulk fill composites in the ART approach — High-viscosity glass-ionomer vs Bulk fill composite to restore shallow and medium depth dentin lesions using the ART approach
  Arms: Shallow and medium depth dentin lesion

SUMMARY:
The present study aims evaluate the oral health conditions of schoolchildren and its relation to growth, development and well-being. Also, it seeks to evaluate different restorative interventions performed at school premises in primary teeth and its impact on the quality of life.

DETAILED DESCRIPTION:
Schoolchildren, aged 6-8 years old, from the six public schools of a deprived suburban area of Brasília, Brazil will be recruited. In the stage 1 of the study, an epidemiological survey of the oral health status and an anthropometric evaluation of the children will be performed. Potential patient for study's stage 2 will be recruited. Quality of life surveys, patterns of oral hygiene and socio-demographic data will be collected.

Children with restorative treatment needs will be included in the study's stage 2. In this second stage, primary molars with deep dentin lesions will be treated according to two techniques for selective excavation of carious dentin: subjective criteria or using an objective criteria (polymer burs). For both groups restorations will be performed using a high-viscosity glass-ionomer. In shallow and medium depth dentin lesions, carious dentin will be excavated using hand instruments only (ART approach) and restored using two materials: a high-viscosity glass-ionomer or a combination of a self-etch adhesive and a bulk fill composite.

All children will be followed up (study's stage 3) to assess efficacy of the restorative interventions and impact of the restorative treatment on children's quality of life and development.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-8 years old;
* Good general health;
* minimum one cavitated dentin carious lesion in a primary molar with sensible asymptomatic pulp.

Exclusion Criteria:

* participating in other study;
* plan to move or not residents;
* systemic disease or general disability;
* expected limited compliance; known allergy to study material; expected exfoliation of primary molars within 18 months.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Success of the restorative procedure | Through study completion, an average of 3 years
  Success of the restorative treatment, not requiring any re-intervention (as endo or extraction). Success will be measured at different time frames.

SECONDARY OUTCOMES:
Survival of the restoration | Through study completion, an average of 3 years
  ART criteria for restoration survival will be used to assess survival of restoration (see Hilgert, 2014)
Quality of life (and change in quality of life) | Baseline and 12months after intervention (change in quality of life)
  Quality of life - Brazilian version of the Early Childhood Oral Health Impact Scale (B-ECOHIS) Questionnaires
Treatment costs | Through study completion, an average of 3 years
  Initial and follow-up treatment costs to allow cost-effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Leandro A Hilgert, PhD, Principal Investigator — University of Brasilia
Locations (1):
- Escolas Públicas do Paranoá / Universidade de Brasília, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricketts D, Lamont T, Innes NP, Kidd E, Clarkson JE. Operative caries management in adults and children. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD003808. doi: 10.1002/14651858.CD003808.pub3. PMID 23543523
- [Background] Hilgert LA, de Amorim RG, Leal SC, Mulder J, Creugers NH, Frencken JE. Is high-viscosity glass-ionomer-cement a successor to amalgam for treating primary molars? Dent Mater. 2014 Oct;30(10):1172-8. doi: 10.1016/j.dental.2014.07.010. Epub 2014 Aug 15. PMID 25132283
- [Background] Schwendicke F, Stolpe M, Innes N. Conventional treatment, Hall Technique or immediate pulpotomy for carious primary molars: a cost-effectiveness analysis. Int Endod J. 2016 Sep;49(9):817-826. doi: 10.1111/iej.12537. Epub 2015 Sep 19. PMID 26331379
- [Background] Schwendicke F, Stangvaltaite L, Holmgren C, Maltz M, Finet M, Elhennawy K, Eriksen I, Kuzmiszyn TC, Kerosuo E, Domejean S. Dentists' attitudes and behaviour regarding deep carious lesion management: a multi-national survey. Clin Oral Investig. 2017 Jan;21(1):191-198. doi: 10.1007/s00784-016-1776-5. Epub 2016 Mar 12. PMID 26971353
- [Background] Schwendicke F, Paris S, Stolpe M. Cost-effectiveness of caries excavations in different risk groups - a micro-simulation study. BMC Oral Health. 2014 Dec 15;14:153. doi: 10.1186/1472-6831-14-153. PMID 25511906
- [Background] De Menezes Abreu DM, Leal SC, Mulder J, Frencken JE. Dental anxiety in 6-7-year-old children treated in accordance with conventional restorative treatment, ART and ultra-conservative treatment protocols. Acta Odontol Scand. 2011 Nov;69(6):410-6. doi: 10.3109/00016357.2011.572561. Epub 2011 Apr 27. PMID 21524172
- [Background] Frencken JE, Leal SC, Navarro MF. Twenty-five-year atraumatic restorative treatment (ART) approach: a comprehensive overview. Clin Oral Investig. 2012 Oct;16(5):1337-46. doi: 10.1007/s00784-012-0783-4. Epub 2012 Jul 24. PMID 22824915
- [Background] de Amorim RG, Figueiredo MJ, Leal SC, Mulder J, Frencken JE. Caries experience in a child population in a deprived area of Brazil, using ICDAS II. Clin Oral Investig. 2012 Apr;16(2):513-20. doi: 10.1007/s00784-011-0528-9. Epub 2011 Mar 8. PMID 21384127
- [Derived] Schwendicke F, Leal S, Schlattmann P, Paris S, Dias Ribeiro AP, Gomes Marques M, Hilgert LA. Selective carious tissue removal using subjective criteria or polymer bur: study protocol for a randomised controlled trial (SelecCT). BMJ Open. 2018 Dec 14;8(12):e022952. doi: 10.1136/bmjopen-2018-022952. PMID 30552261